CLINICAL TRIAL: NCT01863355
Title: Comparison of Analgesic Efficacy and Occurrence of Emesis Among Different Background Infusion and Bolus Administration Regimens of Fentanyl Based Intravenous Patient-controlled Analgesia in Patients After Laparoscopic Assisted Gastrectomy - a Randomized Blind Study -
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0176
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: The Patients With Gastric Cancer Who Are Scheduled to Receive Laparoscopy Assisted Gastrectomy
Keywords: IntravenousPCA, fentanyl, postoperative pain, laparoscopic gastrectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- B0 (Experimental): (basal rate 0cc/hr, bolus 3cc, lockout time 10min)
  Interventions: Drug: B0 group: bolus 0.6mcg/kg without background infusion
- BL (Active Comparator): (basal rate 1cc/hr, bolus 2cc, lockout time 10min)
  Interventions: Drug: BL group: bolus 0.4mcg/kg with background infusion rate 0.2mcg/kg/hr
- BH (Active Comparator): (basal rate 2cc/hr, bolus 1cc, lockout time 10min)
  Interventions: Drug: BH group: bolus 0.2mcg/kg with background infusion rate 0.4mcg/kg/hr

INTERVENTIONS:
Drug: B0 group: bolus 0.6mcg/kg without background infusion
  Other Names: Fentanyl based intraveonus patient controlled analgesia
  Arms: B0
Drug: BL group: bolus 0.4mcg/kg with background infusion rate 0.2mcg/kg/hr
  Other Names: Fentanyl based intraveonus patient controlled analgesia
  Arms: BL
Drug: BH group: bolus 0.2mcg/kg with background infusion rate 0.4mcg/kg/hr
  Other Names: Fentanyl based intraveonus patient controlled analgesia
  Arms: BH

SUMMARY:
Fentanyl based intravenous patient controlled analgesia(PCA)is popular method for postoperative pain control, but information regarding optimal dose of fentanyl in IV PCA is currently lacking. We thus determine appropriate dose of fentanyl (bolus dose and background infusion rate) for effective pain control with minimal side effects such as nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70
* ASA class I and II
* Gastric cancer patients who are scheduled to receive laparoscopic gastrectomy

Exclusion Criteria:

* Cardiovascular disease(uncontrolled hypertension, unstable angina, congestive heart failure, etc.)
* Renal failure
* Liver failure
* Chronic drug or alcohol abuser
* Anti-cancer chemotherapy
* Chronic opioid use
* Use of antiemetics within 24hrs for nausea and vomiting

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain score(VAS) within 48hrs after surgery | Pain socre after surgery 1) within 30min-6hrs, 2) within 6-24hrs, 3) within 24hrs-48hrs
  Pain score after surgery within 48hrs after laparoscopic gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea